CLINICAL TRIAL: NCT00866359
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Followed by an Active-Treatment Extension to Evaluate the Efficacy and Safety of Apremilast(CC-10004) in the Treatment of Behçet Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Apremilast (CC-10004) in the Treatment of Behçet Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-BCT-001; EudraCT#: 2008-002722-11
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Behcet Syndrome
MeSH Terms: conditions — Behcet Syndrome | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. Apremilast (Active Comparator)
  Interventions: Drug: Apremilast (CC-10004)
- B. Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast (CC-10004) — Treatment Phase Days 1-7: Titration from 10 mg BID apremilast tablets arm A (or matching placebo arm B) to 30 mg BID apremilast arm A(or matching placebo arm B) Day 8-84: Maintenance of 30 mg BID apremilast arm A (or matching placebo arm B) Dose reductions to 20 mg BID apremilast arm A (or matching placebo arm B) are permitted.
  Extension Phase All subjects will be given active drug Days 85-91: All placebo subjects from Treatment phase will be dose titrated from 10 mg BID apremilast tablets arm A to 30 mg BID Apremilast.
  Day 92-169: Maintenance of 30 mg BID apremilast arm A or dose reductions to 20 mg BID apremilast arm A (if not previously down titrated)
  Arms: A. Apremilast
Drug: Placebo — Treatment Phase Days 1-7: Titration from 10mg BID matching placebo (arm B) to 30mg BID placebo (arm B) Day 8-84: Maintenance of 30mg BID placebo (arm B). Dose reductions to 20 mg BID matching placebo (arm B) are permitted.
  Extension Phase All subjects will be given active drug Days 85-91: All placebo subjects from Treatment phase will be dose titrated from 10 mg BID apremilast tablets arm A to 30 mg BID Apremilast.
  Day 92-169: Maintenance of 30 mg BID apremilast or dose reductions to 20 mg BID apremilast (if not previously down titrated)
  Arms: B. Placebo Comparator

SUMMARY:
The purpose of this study is to assess whether Apremilast is safe and effective in the treatment of patients with Behcet Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Behçet Disease. At the time of diagnosis, subjects must meet the international study group criteria for Behçet Disease
* Females of childbearing potential (FCBP) must have negative pregnancy tests and agree to use two forms of contraception throughout the study.
* Males must use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP
* Laboratory criteria: Hgb ≥ 9 g/dL, WBC count ≥ 3000 /microL and ≤14,000/microL, platelet count ≥ 100,000 /microL,, serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L), total bilirubin ≤ 2.0 mg/dL, AST and ALT ≤ 1.5 X ULN
* Two or more oral ulcers over the 28 day period before screening, with or without current treatment
* Two or more oral ulcers at the time of randomization (Visit 2, Baseline)

Exclusion Criteria:

* Pregnant or breast feeding
* Any condition which places the subject at risk
* Systemic fungal infection
* History of TB infection within 3 years
* History of recurrent bacterial infection
* Mycobacterium TB as indicated by a positive PPD skin test
* History of incompletely treated Mycobacterium tuberculosis
* Clinically significant chest x-ray abnormality at screening.
* Clinically significant ECG abnormality at screening
* History of HIV infection
* History of congenital or acquired immunodeficiency
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* Antibodies to Hepatitis C at screening
* History of malignancy (except for treated basal-cell skin carcinomas > 3 years prior to screening)
* Any active major organ involvement of Behçet Disease
* Use of concomitant immune modulating therapy or topical corticosteroids.
* Use of ocular corticosteroids
* Use of any investigational medication within 4 weeks prior to randomization or 5 PK/PD half-lives (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (4):
  - Mayo Clinic - Rheumatology and Internal Medicine, Jacksonville, Florida
  - E5, Boston University School of Medicine, Boston, Massachusetts
  - NYU Hospital for Joint Diseases, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Turkey (Türkiye) (3):
  - Eskişehir Osmangazi University, Eskişehir
  - University of Istanbul, Istanbul
  - Selçuk University, Konya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mease PJ, Hatemi G, Paris M, Cheng S, Maes P, Zhang W, Shi R, Flower A, Picard H, Stein Gold L. Apremilast Long-Term Safety Up to 5 Years from 15 Pooled Randomized, Placebo-Controlled Studies of Psoriasis, Psoriatic Arthritis, and Behcet's Syndrome. Am J Clin Dermatol. 2023 Sep;24(5):809-820. doi: 10.1007/s40257-023-00783-7. Epub 2023 Jun 14. PMID 37316690
- [Derived] Hatemi G, Melikoglu M, Tunc R, Korkmaz C, Turgut Ozturk B, Mat C, Merkel PA, Calamia KT, Liu Z, Pineda L, Stevens RM, Yazici H, Yazici Y. Apremilast for Behcet's syndrome--a phase 2, placebo-controlled study. N Engl J Med. 2015 Apr 16;372(16):1510-8. doi: 10.1056/NEJMoa1408684. PMID 25875256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 study sites in Turkey and 3 sites in the United States. The first participant enrolled was enrolled on October 23, 2009 and the last participant enrolled was enrolled on May 08, 2012.
Pre-assignment Details: Eligible participants were randomized 1:1 to receive study drug (apremilast or placebo). Since the incidence and severity of Behçet's Disease differ between males and females, randomization was stratified by gender.
Groups:
- Placebo (Oral) BID: Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets twice daily (BID) in the 12-week placebo-controlled phase.
- Apremilast 30mg (Oral) BID: Treatment Phase (Days 1 to 85): Participants administered to 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
- Placebo/Apremilast 30 mg: Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID started titration doses to reach 30 mg apremilast tablets BID and remained in that dose up to Day 169 in the active treatment extension phase.
- Apremilast 30mg/Apremilast 30mg: Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast BID tablets in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets BID up to Day 169 in the active treatment extension phase.
Period: Treatment Phase (Days 1 to 85)
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Started | 56 | 55 | 0 | 0
Completed | 45 | 50 | 0 | 0
Not Completed | 11 | 5 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Extension Phase (Day 86 to 169)
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Started | 0 | 0 | 45 | 50
Completed | 0 | 0 | 44 | 47
Not Completed | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 3
Period: Observational Follow-Up Phase
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Started | 0 | 0 | 54 (Includes those who entered the follow-up phase from both the placebo controlled or extension phase.) | 54 (Includes those who entered the follow-up phase from both the placebo controlled or extension phase.)
Completed | 0 | 0 | 54 | 54
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population was defined as all randomized participants with at least one oral ulcer evaluation (including the baseline evaluation)
Groups:
- Placebo (Oral) BID: Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets BID in the 12-week placebo-controlled phase.
- Apremilast 30mg (Oral) BID: Treatment Phase (Days 1 to 85): Participants administered 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
- Total: Total of all reporting groups
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.97) | 34.3 (9.11) | 34.5 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 18 | 16 | 34
Duration of Behçet's disease [Mean (Standard Deviation); unit: years] — At the time of diagnosis, participants must meet the 1990 International Study Group criteria for Behçet's Disease. In the absence of other clinical explanations, participants must have: recurrent oral ulceration (apthous or herpetiform) recurring at least 3 times in a 12-month period, plus at least two of the following criteria: 1. Recurrent Genital Ulceration, 2. Eye Lesions, 3. Skin Lesions, 4. Positive Result on Pathergy Testing.
  years | 5.72 (6.084) | 4.92 (3.982) | 5.33 (5.143)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oral Ulcers at Day 85
Description: The number of oral ulcers were counted at each visit and at the end of the treatment period (starting point was at baseline).
Time Frame: Day 85
Population: Intent to Treat (ITT) = all randomized participants with at least one oral ulcer evaluation (including the baseline visit). A Last Observation Carried Forward (LOCF) approach was applied for participants terminated early. If a participant had no post-baseline oral ulcer assessment, the baseline value was carried forward for calculation.
Measure: Least Squares Mean (Standard Error); unit: ulcers/participants
Groups:
- Placebo (Oral) BID: Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets (BID) in the 12-week placebo-controlled phase.
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
ulcers/participants | 2.0 (0.28) | 0.4 (0.28)
Statistical Analysis 1: Comparison: Placebo (Oral) BID vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-2.4 to -0.9] — Based on an analysis of covariance model for the number of ulcers at Day 85, with treatment group and gender as factors and the baseline ulcer number as a covariate

2. Secondary Outcome: Pain of Oral Ulcers as Measured by Visual Analog Scale (VAS) at Day 85
Description: A 100-mm VAS pain scale for oral ulcers was completed by the participant at timepoints specified in the protocol. Each 100-mm VAS was presented to the participant on a single sheet of bond paper. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was measured by ruler and recorded. When responding to a VAS item, participants specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Time Frame: Day 85
Population: The ITT population included all randomized participants with at least one oral ulcer evaluation (including the baseline evaluation). A LOCF approach was applied for participants terminated early from the study. If a participant had no post-baseline oral ulcer assessment, the baseline value was carried forward for calculation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
units on a scale | 36.7 (3.23) | 9.9 (3.30)
Statistical Analysis 1: Comparison: Placebo (Oral) BID vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares mean difference = -26.8, 95% CI 2-sided [-35.5 to -18.0] — Based on an analysis of covariance model for the oral ulcer pain VAS at Day 85, with treatment group and gender as factors and the baseline oral ulcer pain VAS as a covariate

3. Other Pre Specified Outcome: Percentage of Participants Who Were Genital Ulcer-free (Complete Response) at Day 85
Description: The percentage of participants who were genital ulcer-free (complete response: free from active genital ulcers)
Time Frame: Baseline to Day 85
Population: Intent to Treat (ITT) = all randomized participants with at least one genital ulcer at baseline. A Last Observation Carried Forward (LOCF) approach was applied for participants terminated early. If a participant had no post-baseline genital ulcer assessment, the baseline value was carried forward for calculation.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 6 | 10
percentage of participants | 50 | 100

4. Secondary Outcome: Pain of Genital Ulcers as Measured by Visual Analog Scale (VAS) Scores at Day 85
Description: A 100-mm VAS pain scale for genital ulcers was completed by the participant at timepoints specified in the protocol. Each 100-mm VAS was presented to the participant on a single sheet of bond paper. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was measured by ruler and recorded. When responding to a VAS item, participants specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Time Frame: Baseline to Day 85
Population: Not analyzed due to low numbers of genital ulcers; not considered meaningful.
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Area Under the Curve (AUC) for the Number of Oral Ulcers From Day 1 to 85
Description: Area under curve (AUC^85) from Day 1 to Day 85 for the number of oral ulcers per day was determined using the trapezoidal rule and divided by the days between the date of the last observation and baseline. The AUC was determined using the LOCF approach to impute missing values.
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: total AUC (#ulcers*days)
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
total AUC (#ulcers*days) | 157.82 (12.890) | 67.74 (13.267)
Statistical Analysis 1: Comparison: Placebo (Oral) BID vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p < 0.0001, ANCOVA — The last post-baseline observation was carried forward to Day 85 for participants who discontinued the study before Day 85. For participants who did not have Day 85 visit on the targeted date, the total AUC was adjusted by the actual study days; Mean Difference (Final Values) = -90.07, 95% CI 2-sided [-125.32 to -54.82] — Based on an analysis of covariance model for the number of ulcers at Day 85, with treatment group, gender, and interaction of treatment group and gender as factors and the baseline ulcer number as a covariate

6. Secondary Outcome: Area Under the Curve for the Number of Genital Ulcers From Day 1 to 85
Description: Area under curve (AUC^85) from Day 1 to Day 85 for the number of genital ulcers per day was not analyzed.
Time Frame: Day 1 to Day 85
Population: No population analyzed due to small number of participants with genital ulcers; not considered meaningful.
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Area Under the Curve (AUC) for the Number of Oral Plus Genital Ulcers From Day 1 to 85
Description: Area under curve (AUC) from Day 1 to Day 85 (AUC^85) for the number of oral plus genital ulcers per day was determined using the trapezoidal rule and divided by the days between the date of the last observation and baseline. The AUC was determined using the LOCF approach to impute missing values.
Time Frame: Day 1 to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: total AUC (#ulcers*days)
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
total AUC (#ulcers*days) | 193.95 (161.492) | 65.79 (108.037)

8. Secondary Outcome: Sum of the Number Oral Ulcers, Genital Ulcers or Oral Plus Genital Ulcers at Day 85
Description: Sum of the number oral ulcers, genital ulcers or oral plus genital ulcers at Day 85
Time Frame: Day 85
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ulcers/participants
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
Ulcers/participants | 2.3 (0.35) | 0.6 (0.36)
Statistical Analysis 1: Comparison: Placebo (Oral) BID vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.7 to -0.8] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Percentage of Participants Who Were Oral Ulcer-free (Complete Response), or Whose Oral Ulcers Were Reduced by ≥ 50%, (Partial Response)
Description: Comparison of the percentage of participants who were oral ulcer-free (complete response: free from active oral ulcers), or whose oral ulcers were reduced by ≥ 50%, (partial response) between the apremilast-treated and the placebo-treated groups. In this case, partial response also includes complete response.
Time Frame: Baseline and Day 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
percentage of participants
  Complete Response | 28.6 | 70.9
  Partial Response | 50.0 | 89.1
Statistical Analysis 1: Comparison: Placebo (Oral) BID vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Two-sided p-value was based on the CMH test adjusting for gender; adjusted difference (percentage) = 39.1, 95% CI 2-sided [23.6 to 54.5] — Adjusted difference in proportions = weighted average of treatment differences across gender with the CMH weights

10. Secondary Outcome: Change From Baseline in the Disease Activity as Measured by BD Current Activity Form/Index Score on Day 85
Description: The Behçet's Disease Current Activity Index consists of three component scores, a participant's perception of disease activity, a clinician's overall perception of disease activity and a Behçet's Disease Current Activity Index Score. The score ranges from 0 to 12. A higher score indicates higher level of disease activity (worsening) and a negative change from baseline indicates improvement.
Time Frame: Day 1 to Day 85 or to early termination visit
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets BID in the 12-week placebo-controlled phase.
Arm/Group | Placebo | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 55 | 54
units on a scale | -0.1 (0.22) | -1.2 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30mg (Oral) BID; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.7 to -0.5] — Based on an Ancova model for change from baseline with treatment group, gender and interaction of treatment group and gender as factors and the baseline value as a covariate

11. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAE) During the Placebo Controlled Treatment Phase
Description: A Treatment Emergent Adverse Event (TEAE) was defined as any AE occurring or worsening on or after the first treatment of any study drug, and within 28 days after the last dose of the last study drug. A treatment related toxicity was considered by the investigator to be not suspected or suspected. Severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on a 1-5 scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5=Death related to AE.
Time Frame: Day 1 to Day 85; maximum exposure to study drug was 13 weeks during treatment phase
Population: Safety Population defined as all participants who were randomized and received at least 1 dose of Investigational Product.
Measure: Number; unit: participants
Groups:
- Apremilast 30mg (Oral) BID: Treatment Phase (Days 1 to 85): Participants randomized to 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
participants
  Any TEAE | 50 | 49
  Any drug related TEAE | 24 | 30
  Any severe TEAE | 5 | 5
  Any serious TEAE | 3 | 2
  Any serious drug related TEAE | 1 | 0
  Any TEAE leading to drug interruption | 0 | 1
  Any TEAE leading to drug withdrawal | 5 | 4

12. Secondary Outcome: Number of New Manifestations of Behçet's Disease or Flare During the Placebo Controlled Treatment Phase
Description: A flare was defined as the development of new manifestations of BD or worsening of existing disease, meeting the following criteria:
  1. Organ involvement: any major organ involvement (eg, central nervous system, gastrointestinal tract);
  2. Oral/genital ulcers: ≥ 100% increase in the number of oral or genital ulcers from Day 1 or a minimum increase of 3 in the number of oral or genital ulcers, whichever is greater;
  3. Arthritis: ≥ 50% increase in the number of swollen joints, or a minimum increase of 3 swollen joints, whichever is greater;
  4. Skin lesions (non-oral/genital ulcers): ≥ 50% increase in the total score of the Physician's Global Assessment of Skin Lesions, or a minimum increase of 2 in the total score of the Physician's Global Assessment of Skin Lesions, whichever is greater'
  5. New onset or worsening of existing Behçet Disease-related inflammatory eye disease requiring initiation of immunosuppressive therapy (uveitis).
Time Frame: Day 1 to Day 85
Population: Safety population included all participants who were randomized and received at least 1 dose of Investigational Product.
Measure: Number; unit: participants
Arm/Group | Placebo (Oral) BID | Apremilast 30mg (Oral) BID
Number analyzed (Participants) | 56 | 55
participants
  Participants who had disease flare | 27 | 12
  Participants with new onset or worsening uveitis | 3 | 0

13. Secondary Outcome: Number of Oral Ulcers at Day 169
Description: The number of oral ulcers were counted at Day 169 in reference to the participants' first day of active treatment (Day 1 or Day 85).
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ulcers/participant
Groups:
- Apremilast 30 mg /Apremilast 30mg BID (Oral): Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets BID in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast BID up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30 mg /Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 45 | 49
ulcers/participant | 0.4 (1.31) | 0.6 (1.27)

14. Secondary Outcome: Pain of Oral Ulcers as Measured by VAS (VAS Score) at Day 169
Description: as for outcome 2
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 30 mg /Apremilast 30mg BID (Oral): Extension Phase (Days 86 to 169): Participants initially administered to receive 30 mg apremilast tablets BID in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast BID up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30 mg /Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 45 | 47
units on a scale | 9.6 (21.13) | 9.7 (20.33)

15. Other Pre Specified Outcome: Percentage of Participants Who Were Genital Ulcer-free (Complete Response) at Day 169
Description: The percentage of participants who were genital ulcer-free (complete response: free from active genital ulcers)
Time Frame: Day 1 to Day 169
Population: Intent to Treat (ITT) = all randomized participants with at least one genital ulcer at baseline visit. A Last Observation Carried Forward (LOCF) approach was applied for participants terminated early. If a participant had no post-baseline genital ulcer assessment, the baseline value was carried forward for calculation.
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 30mg/Apremilast 30mg: Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Number analyzed (Participants) | 6 | 10
percentage of participants | 66.7 | 100

16. Secondary Outcome: Pain of Genital Ulcers as Measured by Visual Analog Scale (VAS) at Day 169
Description: as for outcome 4
Time Frame: Day 1 to Day 169
Population: Not analyzed due to low numbers of genital ulcers; not considered meaningful.
Groups:
- Placebo BID/Apremilast 30 BID (Oral): Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID started titration doses to reach 30 mg apremilast tablets BID and remained in that dose up to Day 169 in the active treatment extension phase .
- Apremilast 30 mg BID/Apremilast 30mg BID (Oral): Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo BID/Apremilast 30 BID (Oral) | Apremilast 30 mg BID/Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Behçet's Disease (BD) Current Activity Index Form Score at Day 169
Description: as for outcome 10
Time Frame: Day 169
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 30mg/Apremilast 30mg: Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID were titrated to 30 mg apremilast tablets BID up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Number analyzed (Participants) | 45 | 49
units on a scale | 1.4 (1.18) | 1.6 (1.62)

18. Secondary Outcome: Number of New Manifestations of Behçet's Disease or Flare That Were Not Present at Day 1
Description: A flare was defined as the development of new manifestations of BD or worsening of existing disease, meeting the following criteria:
  1. Organ involvement: any major organ involvement (eg, central nervous system, gastrointestinal tract);
  2. Oral/genital ulcers: ≥ 100% increase in the number of oral or genital ulcers from Day 1 or a minimum increase of 3 in the number of oral or genital ulcers, whichever is greater;
  3. Arthritis: ≥ 50% increase in the number of swollen joints, or a minimum increase of 3 swollen joints, whichever is greater;
  4. Skin lesions (non-oral/genital ulcers): ≥ 50% increase in the total score of the Physician's Global Assessment of Skin Lesions, or a minimum increase of 2 in the total score of the Physician's Global Assessment of Skin Lesions, whichever is greater;
  5. New onset or worsening of existing Behçet Disease-related inflammatory eye disease requiring initiation of immunosuppressive therapy (uveitis).
Time Frame: Day 1 to Day 169
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Apremilast 30mg/Apremilast 30mg: Treatment and Extension Phases (Days 1 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Number analyzed (Participants) | 45 | 55
participants
  Participants who experienced a disease flare | 15 | 19
  Participants with new onset or worsening uveitis | 1 | 2

19. Secondary Outcome: Number of Oral Ulcers at Day 197
Description: as for outcome 1
Time Frame: Day 197
Population: Includes participants who entered the Observational Follow-up Phase from either the Treatment Phase or the Extension Phase
Measure: Mean (Standard Deviation); unit: ulcers/participants
Groups:
- Placebo/Apremilast 30 mg: Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets twice daily (BID) in the 12-week placebo-controlled phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID started titration doses to reach 30 mg apremilast tablets BID and remained in that dose up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
- Apremilast 30 mg /Apremilast 30mg BID (Oral): Treatment Phase (Days 1 to 85): Participants administered 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30 mg /Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 54 | 54
ulcers/participants | 1.6 (1.78) | 1.7 (2.06)

20. Secondary Outcome: Pain of Oral Ulcers as Measured by VAS (VAS Score) at Day 197
Description: as for outcome 2
Time Frame: Day 197
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30 mg /Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 54 | 54
units on a scale | 21.0 (22.26) | 27.2 (28.71)

21. Other Pre Specified Outcome: Percentage of Participants Who Were Genital Ulcer-free (Complete Response)
Description: The percentage of participants who were genital ulcer-free (complete response: free from active genital ulcers)
Time Frame: Day 1 to Day 197
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Groups:
- Apremilast 30mg/Apremilast 30mg: Treatment Phase (Days 1 to 85): Participants administered 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30mg/Apremilast 30mg
Number analyzed (Participants) | 6 | 10
percentage of participants | 100 | 100

22. Secondary Outcome: Pain of Genital Ulcers as Measured by Visual Analog Scale (VAS) at Day 197
Description: as for outcome 4
Time Frame: Day 1 to Day 197
Population: Not analyzed due to low numbers of genital ulcers; not considered meaningful.
Groups:
- Placebo BID/Apremilast 30 BID (Oral): Treatment Phase (Days 1 to 85): Participants administered identically matching placebo tablets twice daily (BID) in the 12-week placebo-controlled phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID started titration doses to reach 30 mg apremilast tablets BID and remained in that dose up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
- Apremilast 30 mg BID/Apremilast 30mg BID (Oral): Treatment Phase (Days 1 to 85): Participants administered 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
Arm/Group | Placebo BID/Apremilast 30 BID (Oral) | Apremilast 30 mg BID/Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Change From Baseline in the Disease Activity as Measured by BD Current Activity Form/Index Score on Day 197
Description: as for outcome 10
Time Frame: Day 1 to Day 197
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Apremilast 30 mg/Apremilast 30mg BID: Treatment Phase (Days 1 to 85): Participants administered 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase.
  Extension Phase (Days 86 to 169): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled treatment phase continued to receive 30 mg apremilast tablets twice daily up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
Arm/Group | Placebo/Apremilast 30 mg | Apremilast 30 mg/Apremilast 30mg BID
Number analyzed (Participants) | 53 | 53
units on a scale | -0.6 (1.28) | -1.2 (1.65)

24. Secondary Outcome: Summary of Treatment Emergent Adverse Events During the Active Treatment-Extension Phase
Description: A Treatment Emergent Adverse Event (TEAE) is as any AE occurring or worsening on or after the first treatment of any study drug, and within 28 days after the last dose of the last study drug. A treatment related toxicity was considered by the investigator to be not suspected or suspected. Severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on a 1-5 scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5=Death related to AE.
Time Frame: Day 1 to Day 197; maximum exposure was 25.1 weeks
Population: Safety analyses for the apremilast-exposure period was based on the apremilast participants as treated (AAT) Population, and included those who were randomized (at the randomization visit) or switched (at the Day 85 visit) to apremilast 30 mg BID, and received at least one dose of apremilast after the initial randomization or switch to 30 mg BID.
Measure: Number; unit: particpants
Groups:
- Placebo BID/Apremilast 30 BID (Oral): Extension Phase (Days 86 to 169): Participants initially randomized to placebo BID started titration doses to reach 30 mg apremilast tablets BID and remained in that dose up to Day 169 in the active treatment extension phase.
  Day 197 includes those who entered the follow-up phase from both the placebo controlled or extension phase.
Arm/Group | Placebo BID/Apremilast 30 BID (Oral) | Apremilast 30 mg BID/Apremilast 30mg BID (Oral)
Number analyzed (Participants) | 45 | 55
particpants
  Any TEAE | 39 | 50
  Any drug related TEAE | 20 | 33
  Any severe TEAE | 1 | 11
  Any serious TEAE | 1 | 5
  Any serious drug related TEAE | 0 | 1
  TEAE leading to drug interuption | 0 | 1
  TEAE leading to drug withdrawal | 1 | 7

ADVERSE EVENTS:
Time Frame: Days 1 to Day 197 visit; maximum exposure to study drug was 25.1 weeks. From Day 1 (first dose) through the end of the follow up period up to 28 days after the last dose of study drug.
Description: 108 participants were part of the follow-up phase (had prematurely discontinued therapy during the placebo (PBO)-controlled phase but had completed PBO-controlled phase and prematurely discontinued therapy during the extension phase. Those who prematurely discontinued therapy during the PBO-controlled phase did not participate the extension phase
Groups:
- Week 12: Placebo BID: Participants randomized to placebo tablets twice daily during the placebo-controlled phase. Includes data through Week 12 for all participants randomized to placebo.
- Week 12: Apremilast 30 mg BID: Participants randomized to 30 mg Apremilast tablets BID during the 12-week placebo-controlled treatment phase. Includes data through Week 12 for all participants randomized to 30mg Apremilast BID.
- Week 24: Apremilast 30 mg BID: Participants who received 30 mg apremilast, regardless of when the apremilast exposure started (at Week 0, or 12), up until Week 24. Includes data through Week 24 for participants who were treated with Apremilast started at Week 0 and data from Week 12 through Week 24 for participants who were treated with Apremilast started at Week 12.
Arm/Group | Week 12: Placebo BID | Week 12: Apremilast 30 mg BID | Week 24: Apremilast 30 mg BID
Serious Adverse Events (participants affected / at risk) | 3/56 | 2/55 | 6/100
Other Adverse Events (participants affected / at risk) | 48/56 | 47/55 | 82/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Week 12: Placebo BID (N=56) | Week 12: Apremilast 30 mg BID (N=55) | Week 24: Apremilast 30 mg BID (N=100)
Behçet's Syndrome (Immune system disorders) | 2 | 0 | 3
Diplegia (Nervous system disorders) | 0 | 1 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Pyrexia (Gastrointestinal disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Week 12: Placebo BID (N=56) | Week 12: Apremilast 30 mg BID (N=55) | Week 24: Apremilast 30 mg BID (N=100)
Influenza (Infections and infestations) | 1 | 3 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 2 | 6
Oral Herpes (Infections and infestations) | 4 | 2 | 4
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 6
Behçet's Syndrome (Immune system disorders) | 25 | 12 | 35
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 5 | 5
Headache (Nervous system disorders) | 25 | 26 | 41
Hypoaesthesia (Nervous system disorders) | 1 | 4 | 4
Dizziness (Nervous system disorders) | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6
Nausea (Gastrointestinal disorders) | 10 | 22 | 36
Diarrhoea (Gastrointestinal disorders) | 2 | 12 | 20
Abdominal Pain (Gastrointestinal disorders) | 7 | 8 | 11
Vomiting (Gastrointestinal disorders) | 1 | 9 | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 3 | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 6 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Asthenia (General disorders) | 2 | 5 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Insomnia (Psychiatric disorders) | 0 | 0 | 5
Depression (Psychiatric disorders) | 0 | 0 | 5

LIMITATIONS AND CAVEATS:
Planned sample size not reached; slow enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 45 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential data before submission or defer publication to permit patent applications.